CLINICAL TRIAL: NCT00544232
Title: Randomized Comparison of a Preoperative, Dose-Intensified, Interval-Shortened, Sequential Chemotherapy With Epirubicin, Paclitaxel and CMF ± Darbepoetin Alfa Versus a Preoperative, Sequential Chemotherapy With Epirubicin and Cyclophosphamide Followed by Paclitaxel in Standard Dosage ± Darbepoetin Alfa in Patients With Primary Breast Cancer
Brief Title: Preoperative Epirubicin Paclitaxel Aranesp Study (PREPARE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Pharmacia (Industry); Amgen (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 49
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; neoadjuvant therapy; pCR rates
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Paclitaxel; Cyclophosphamide; Methotrexate; Fluorouracil; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- epirubicin, paclitaxel and CMF +/- darbepoetin (Experimental): Epirubicin (90 mg/m2) d1, q21d - 4× / cyclophosphamide (600 mg/m2) d1, q21d - 4× followed by paclitaxel (175 mg/m2) d1, q21d - 4×
  +/- Darbepoetin alfa 1 × 4.5 μg/kg of body weight every two weeks with the start of the first epirubicin dose (day 1) to 14 days after the last dose of paclitaxel
  Interventions: Drug: Epirubicin, paclitaxel, cyclophosphamide, Methotrexate, 5 FU, darbepoetin alfa
- EC followed by paclitaxel +/- darbepoetin (Experimental): Epirubicin (150 mg/m2) d1, q14d - 3× followed by paclitaxel (225 mg/m2) d1, q14d - 3×, followed by CMF d1/d8, q28d - 3× Obligatory pegfilgratim 6 mg, subcutaneous injection on day 2 after epirubicin and/or paclitaxel and secondary prophylactic dose after CMF
  +/- Darbepoetin alfa 1 × 4.5 μg/kg of body weight every two weeks with the start of the first dose of epirubicin (day 1) until 14 days after the last dose of CMF
  Interventions: Drug: Epirubicin, Cyclophosphamide, Paclitaxel, dabepoetin alfa

INTERVENTIONS:
Drug: Epirubicin, paclitaxel, cyclophosphamide, Methotrexate, 5 FU, darbepoetin alfa — Epirubicin (90 mg/m2) d1, q21d - 4× / cyclophosphamide (600 mg/m2) d1, q21d - 4× followed by paclitaxel (175 mg/m2) d1, q21d - 4×
  +/- Darbepoetin alfa 1 × 4.5 μg/kg of body weight every two weeks with the start of the first epirubicin dose (day 1) to 14 days after the last dose of paclitaxel
  Arms: epirubicin, paclitaxel and CMF +/- darbepoetin
Drug: Epirubicin, Cyclophosphamide, Paclitaxel, dabepoetin alfa — Epirubicin (150 mg/m2) d1, q14d - 3× followed by paclitaxel (225 mg/m2) d1, q14d - 3×, followed by CMF d1/d8, q28d - 3× Obligatory pegfilgratim 6 mg, subcutaneous injection on day 2 after epirubicin and/or paclitaxel and secondary prophylactic dose after CMF
  +/- Darbepoetin alfa 1 × 4.5 μg/kg of body weight every two weeks with the start of the first dose of epirubicin (day 1) until 14 days after the last dose of CMF
  Arms: EC followed by paclitaxel +/- darbepoetin

SUMMARY:
The present clinical trial will investigate the efficacy of a sequential interval-shortened and dose-intensified preoperative use of epirubicin, paclitaxel and CMF with preoperative sequential administration of epirubicin and cyclophosphamide followed by paclitaxel in breast cancer. In addition, the influence of darbepoetin alfa on the response rate and quality of life is to be investigated in both treatment arms.

DETAILED DESCRIPTION:
Arm A: Sequential treatment in standard doses with Epirubicin (90 mg/m2)/cyclophosphamide (600 mg/m2) d1, q21d - 4× followed by paclitaxel (175 mg/m2) d1, q21d - 4×.

Pegfilgratim should be used as secondary preventive after febrile neutropenia in the standard arm of the study, or in exceptional cases also after severe febrile neutropenia necessitating postponement of the treatment by more than one week ± Darbepoetin alfa 1 × 4.5 µg/kg of body weight every two weeks with the start of the first epirubicin dose (day 1) until 14 days after the last dose of paclitaxel Daily oral intake of 200 mg iron unless there complications occur with taking iron

Arm B: sequential dose-intensified, interval-shortened treatment with Epirubicin (150 mg/m2) d1, q14d - 3× followed by paclitaxel (225 mg/m2) d1, q14d - 3×, followed by CMF (600/40/600 mg/m2) d1/d8, q28d - 3× Obligatory pegfilgratim 6 mg after epirubicin and/or paclitaxel: subcutaneous injection on day 2. After CMF pegfilgrastim should be used as a secondary preventive measure

± Darbepoetin alfa 1 × 4.5 µg/kg of body weight every two weeks with the start of the first dose of epirubicin (day 1) until 14 days after the last dose of CMF Daily oral dose of 200 mg iron unless complications occur in taking iron.

Primary goal: Determining the relapse-free survival time and overall survival after dose-intensified sequential preoperative chemotherapy including anthracycline and taxan and/or after preoperative chemotherapy including anthracycline followed by taxan in a standard dose

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer: at least three fast biopsies.
* Primary tumor ≥2 cm acc. to clinical measurement or manifestation of an inflammatory breast cancer.
* No systemic metastasis, exclusion by chest x-ray, sonogram of the upper abdomen and skeletal scintiscan.
* Age ≥18 years and ≤65 years.
* ECOG < 2/WHO 0-1
* Adequate organ function defined as SGOT and bilirubin ≤ 1.5× upper limit WBC ≥ 3000 /µL Neutrophils ≥ 1000 /µL Platelets ≥ 100,000 /µL Serum creatinine < 2.0 mg/dL
* Unremarkable heart echo
* No florid hepatitis
* Written consent to participate in the treatment optimization protocol

Exclusion Criteria:

* Multicentricity in various quadrants (contact the study office)
* Known allergy to E. coli-produced medication
* Known allergy to medication containing cremophor (e.g., cyclosporin A)
* Patients receiving immunosuppressant therapy
* Lack of consent after informing the patient
* Lack of willingness to keep and disclose personal medical data as part of the study
* Pregnancy, nursing
* Secondary malignancy, excluding basalioma of the skin or carcinoma in situ of the cervix that has received curative therapy
* Pre-existing treatment-resistant cardiac disease, coronary heart disease, arrhythmias, cardiac insufficiency
* Patients with uncontrolled hypertension (diastolic >95 mmHg)
* A history of convulsions
* Known hypersensitivity to darbepoetin alfa or any of its other ingredients or a known hypersensitivity to r-HuEPO

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2002-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival time and overall survival | 2007

CONTACTS AND LOCATIONS:
Overall Officials: M. Untch, MD, Principal Investigator — Clinic of the Ludwig-Maximilian-University, München

REFERENCES:
- [Result] Untch M, Fasching PA, Konecny GE, von Koch F, Conrad U, Fett W, Kurzeder C, Luck HJ, Stickeler E, Urbaczyk H, Liedtke B, Salat C, Harbeck N, Muller V, Schmidt M, Hasmuller S, Lenhard M, Schuster T, Nekljudova V, Lebeau A, Loibl S, von Minckwitz G; Arbeitsgemeinschaft Gynakologische Onkologie PREPARE investigators. PREPARE trial: a randomized phase III trial comparing preoperative, dose-dense, dose-intensified chemotherapy with epirubicin, paclitaxel and CMF versus a standard-dosed epirubicin/cyclophosphamide followed by paclitaxel +/- darbepoetin alfa in primary breast cancer--results at the time of surgery. Ann Oncol. 2011 Sep;22(9):1988-1998. doi: 10.1093/annonc/mdq709. Epub 2011 Mar 8. PMID 21385882
- [Result] Untch M, von Minckwitz G, Konecny GE, Conrad U, Fett W, Kurzeder C, Luck HJ, Stickeler E, Urbaczyk H, Liedtke B, Beckmann MW, Salat C, Harbeck N, Muller V, Schmidt M, Hasmuller S, Lenhard M, Nekljudova V, Lebeau A, Loibl S, Fasching PA; Arbeitsgemeinschaft Gynakologische Onkologie PREPARE investigators. PREPARE trial: a randomized phase III trial comparing preoperative, dose-dense, dose-intensified chemotherapy with epirubicin, paclitaxel, and CMF versus a standard-dosed epirubicin-cyclophosphamide followed by paclitaxel with or without darbepoetin alfa in primary breast cancer--outcome on prognosis. Ann Oncol. 2011 Sep;22(9):1999-2006. doi: 10.1093/annonc/mdq713. Epub 2011 Mar 7. PMID 21382868
- [Derived] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812